CLINICAL TRIAL: NCT04279106
Title: "Effect of Single Rinsing With Three Different Types of Mouthwash on VSC Levels in Morning Breath; Randomized Clinical Trial, Double-blind Cross-sectional Study"
Brief Title: Effect of Single Rinsing With Three Different Types of Mouthwash on VSC Levels in Morning Breath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Enrico Marchetti, Adjunct Professor, University of L'Aquila
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: RCT-01-2020
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Halitosis
Keywords: Morning bad breath; Halitosis; OralChroma; mouthwash
MeSH Terms: conditions — Halitosis | interventions — Ethanol; Listerine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0.05%chlorhexidine mouthwash (Experimental): All subjects were instructed to rinse once a day, in the morning, with 15 ml solution for 60 seconds, after which they expectorated. Subsequent rinsing with water was not allowed.
  Interventions: Procedure: 0.05%chlorhexidine mouthwash
- 0.05% sodium fluoride mouthwash (Active Comparator): All subjects were instructed to rinse once a day, in the morning, with 15 ml solution for 60 seconds, after which they expectorated. Subsequent rinsing with water was not allowed.
  Interventions: Procedure: 0.05% sodium fluoride mouthwash
- alcohol free essential oils mouthwash (Active Comparator): All subjects were instructed to rinse once a day, in the morning, with 15 ml solution for 60 seconds, after which they expectorated. Subsequent rinsing with water was not allowed.
  Interventions: Procedure: alcohol free essential oils mouthwash
- Placebo (Placebo Comparator): All subjects were instructed to rinse once a day, in the morning, with 15 ml solution for 60 seconds, after which they expectorated. Subsequent rinsing with water was not allowed.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: 0.05%chlorhexidine mouthwash — All subjects were instructed to rinse once a day, in the morning, with 15 ml solution for 60 seconds, after which they expectorated. Subsequent rinsing with water was not allowed.
  Other Names: Mentadent professional 0.05%chlorhexidine. MIROMED Srl
  Arms: 0.05%chlorhexidine mouthwash
Procedure: 0.05% sodium fluoride mouthwash — All subjects were instructed to rinse once a day, in the morning, with 15 ml solution for 60 seconds, after which they expectorated. Subsequent rinsing with water was not allowed.
  Other Names: CB12®.Mylan N.V.
  Arms: 0.05% sodium fluoride mouthwash
Procedure: alcohol free essential oils mouthwash — All subjects were instructed to rinse once a day, in the morning, with 15 ml solution for 60 seconds, after which they expectorated. Subsequent rinsing with water was not allowed.
  Other Names: Listerine, Johnson & Johnson Consumer Inc.
  Arms: alcohol free essential oils mouthwash
Procedure: Placebo — All subjects were instructed to rinse once a day, in the morning, with 15 ml solution for 60 seconds, after which they expectorated. Subsequent rinsing with water was not allowed.
  Arms: Placebo

SUMMARY:
Morning bad breath (MBB) is often an enduring upset; this double blind, crossover, randomized study aimed to evaluate the bad breath-suppressing of 3 commercially available mouth rinses (Mentadent Professional® 0.05%chlorhexidine (MPc), Meridol® Halitosis (MH) and CB12®) and a placebo on morning halitosis during a washout period of 1 week.

DETAILED DESCRIPTION:
The study was designed as a double-masked, four-group, randomized, crossover clinical trial.

The volunteers were randomly assigned. Randomization was performed using computer generated random numbers. The allocation of active or control solutions was undertaken by a person not directly involved in the research project. No changes to methods after trial commencement (such as eligibility criteria) were performed.

Participants Thirty-six nondental student volunteers (17 women and 15 men; age range 34-22 years old; mean age 27,7) participated in the study. The subjects were recruited through advertisements. All of the candidates were screened for suitability by the research team. The selection criteria were: Good general health condition, dentition with ≥20 evaluable teeth (minimum of five teeth per quadrant), no oral lesions, no severe periodontal problems (no probing depth ≥5 mm or attachment loss >2 mm), and no removable prostheses or orthodontic bands or appliances. Persons allergic to several mouthwash components were excluded from the study. All eligible volunteers were given oral and written information about the products and the purpose of the study and were asked to sign an informed consent form. The study was conducted from 3 September 2018 to 10 December 2019 in the Division of Periodontology, University of L'Aquila.

During the first information meeting, at each participant was given the mouthwash samples to be tested and a sealed envelope in which the sequence to follow was specified. The sequence also included the use of a placebo. The subjects were asked not to change their eating habits, but to refrain from taking halogen substances on the evenings prior the evaluations.

About 12 hours before the analysis, the participants, refraining from oral hygiene practices, performed a 30-second rinse, followed by a gargle. They also committed themselves not to take food or drinks, not to brush their teeth, not to smoke and not to use cosmetics (their fragrances could have disturbed the operator's perception of odours), between this practice and the evaluation.

The following morning the values of hydrogen sulphide, methyl mercaptan and dimethyl sulphide were measured and the values of the Rosenberg scale (0. Absence of odor;1. Barely perceptible odor;2. Slight but clearly perceptible odor;3. Moderate odour; 4. Very annoying smell; 5. Extremely bad smell) and the Winkel index (0. Absence of patina;1. Slight presence of patina; 2. Considerable presence of patina) were assigned. The assessment of morning halitosis was carried out through organoleptic measurement with a lingual patina supervision and with the aid of a dedicated device, the Oral Chroma.

ELIGIBILITY:
Inclusion Criteria:

* age between 20 and 50 years old

Exclusion Criteria:

* oral lesions
* severe periodontal problems (probing depth ≥5 mm or attachment loss >2 mm)
* removable prostheses or orthodontic bands/ or appliances
* Subjects allergic to several mouthrinse

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Level of VSCs | 1Day
  The detection of halitosis with gas chromatography, which allows to obtain the exact values of VSCs present in the exhaled air, was performed trough the OralChroma. For the practical test, patients were asked to breathe through the nose for a couple of minutes, after inserting a 10 ml disposable syringe deprived of the needle in the oral cavity

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Marzo, DMD, Study Chair — University of L'Aquila
Locations (1):
- University of L'Aquila, Division of Periodontology, L’Aquila, AQ, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marchetti E, Casalena F, Capestro A, Tecco S, Mattei A, Marzo G. Efficacy of two mouthwashes on 3-day supragingival plaque regrowth: a randomized crossover clinical trial. Int J Dent Hyg. 2017 Feb;15(1):73-80. doi: 10.1111/idh.12185. Epub 2015 Nov 2. PMID 26522915
- [Background] Marchetti E, Mummolo S, Di Mattia J, Casalena F, Di Martino S, Mattei A, Marzo G. Efficacy of essential oil mouthwash with and without alcohol: a 3-day plaque accumulation model. Trials. 2011 Dec 15;12:262. doi: 10.1186/1745-6215-12-262. PMID 22171999
- [Background] Mendes L, Coimbra J, Pereira AL, Resende M, Pinto MG. Comparative effect of a new mouthrinse containing chlorhexidine, triclosan and zinc on volatile sulphur compounds: a randomized, crossover, double-blind study. Int J Dent Hyg. 2016 Aug;14(3):202-8. doi: 10.1111/idh.12132. Epub 2015 Feb 26. PMID 25727335
- [Background] van Steenberghe D, Avontroodt P, Peeters W, Pauwels M, Coucke W, Lijnen A, Quirynen M. Effect of different mouthrinses on morning breath. J Periodontol. 2001 Sep;72(9):1183-91. doi: 10.1902/jop.2000.72.9.1183. PMID 11577950